CLINICAL TRIAL: NCT02146183
Title: Compositions Comprising a Steviol Glycoside for Use in Restoring Muscle Glycogen by Increasing the Rate of Glycogen Re-synthesis in Muscles
Brief Title: Steviol Glycoside for Use in Restoring Muscle Glycogen by Increasing the Rate of Glycogen Re-synthesis in Muscles
Acronym: steviagly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Per Bendix Jeppesen (Other)
Collaborators: University of Aarhus (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Per Bendix Jeppesen, Associate Prof, PhD, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Aarhus University
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Glycogen Depletion
Keywords: Stevio glycosides; sport; glycogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo / Corn starch (Placebo Comparator): Carbohydrate-containing composition that comprises 2 g carbohydrate per kg of body weight. This composition will be 500 mg placebo starch corn.
  Interventions: Dietary Supplement: Placebo Corn Starch
- Carbohydrate steviol glycosides (Active Comparator): 500 mg steviol glycosides.
  Interventions: Dietary Supplement: Carbohydrate steviol glycosides

INTERVENTIONS:
Dietary Supplement: Carbohydrate steviol glycosides — To investigate if intake of stevioside in addition to a carbohydrate-containing composition after work related depletion of muscle glycogen will increase the rate of glycogen re-synthesis as compared with intake of the carbohydrate-containing composition alone.
  Arms: Carbohydrate steviol glycosides
Dietary Supplement: Placebo Corn Starch — 500 mg/day
  Arms: placebo / Corn starch

SUMMARY:
The aim of this experiment is to investigate if intake of stevioside in addition to a carbohydrate-containing composition after work related depletion of muscle glycogen will increase the rate of glycogen re-synthesis as compared with intake of the carbohydrate-containing composition alone.

DETAILED DESCRIPTION:
Test subjects Healthy and well trained male subjects will be selected for the study. The subjects will be completing the test procedure twice, on two separate days at least 7 days apart in a crossover design, where intervention - i.e. addition of stevioside to the restitution meal - is blinded and randomised for both the test subjects and the scientific staff.

Inclusion criteria:

Well trained, healthy exhaustive trained males, age 18 to 40.

Exclusion criteria:

Persons suffering of a metabolic disease, which is related to the carbohydrate metabolism, such as diabetes type 1 or 2, insulin resistance and the like, cannot be included in the test. Also persons, who are prescribed a medical drug or diet supplement that could affect the carbohydrate metabolism, will be excluded from the study. Finally persons that are not capable of completing the fasting period or the test design will be excluded from the study.

Before testing Before testing the VO2-max and maximal pulse will be determined for each test subject. The results of this test will be used for determination of the working load for each test subject during the test.

The test will be performed for at least 72 hours before the bicycling test is commenced.

Experimental design:

The bicycling test is designed as a working session having the purpose of completely depleting the muscle glycogen storage of the working muscles. The depletion of muscle glycogen will be further facilitated by a twelve hours fasting period prior to commencement of the bicycling test.

The test persons will be completing the test twice on two separate days at least 7 days apart in a crossover design, where the intervention - i.e. the additional intake of stevioside together with the carbohydrate-containing composition during the bicycling work - is blinded and randomised for both the test subjects and the scientific staff.

During the working session the test subjects will be exercising for 2 hours on a bicycle ergometer at 65-75% of VO2-max. Afterwards these two hours of bicycling exercise, the persons will be performing a number of one minute intervals at maximum workload. Every interval will be followed by a one minute break, where the subjects pedal at low intensity of own choice. This interval exercise will be continued until the test subject's plasma glucose is below 3.89 mmol/l. This value is selected to ensure that the glycogen storage in the liver is depleted to identical extent in each test.

Immediately after the working session the test subject will be given a carbohydrate-containing composition that comprises 2 g carbohydrate per kg of body weight. Also 2 hours after completion of the working session the test persons will be given a carbohydrate-containing composition that comprises 2 g carbohydrate per kg of body weight. These compositions will be added either 500 mg stevioside or placebo (starch corn).

Tissue and blood samples Before the working session will be commenced blood samples will be collected together with muscle biopsies in order to determine the content of plasma glucose, plasma insulin, and muscle glycogen before commencement of the bicycling workload. Further blood samples will be collected at 0, 30, 60, 90, 120, 150, 180, 210 and 240 minutes after completion of the working session, and further muscle biopsies will be collected at 0, 120 and 240 minutes after completion of the working session.

After collection the blood samples will be centrifuged and the serum will be stored at -20°C. Parameters that will be evaluated in the blood samples will be content of glucose, insulin, glycagon, kreatine kinase, lactate dehydrogenase and myoglobin.

After collection of the muscle biopsies the samples will be stored under liquid nitrogen. The parameter evaluated in the muscles biopsies will be glycogen.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:
* Healthy and well trained, sporty exhaustive trained males, age 18 to 40 years old.

Exclusion Criteria:

* Persons suffering of a metabolic disease, which is related to the carbohydrate metabolism, such as diabetes type 1 or 2, insulin resistance and the like, cannot be included in the test. Also persons, who are prescribed a medical drug or diet supplement that could affect the carbohydrate metabolism, will be excluded from the study. Finally persons that are not capable of completing the fasting period or the test design will be excluded from the study.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-02 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Effects on glycogen re-synthesis | 2 weeks
  During the working session the test subjects will be exercising for 2 hours on a bicycle ergometer at 65-75% of VO2-max.
  Immediately after the working session the test subject will be given a carbohydrate-containing composition that comprises 2 g carbohydrate per kg of body weight. Also 2 hours after completion of the working session the test persons will be given a carbohydrate-containing composition that comprises 2 g carbohydrate per kg of body weight. These compositions will be added either 500 mg stevioside or placebo (starch corn).
  After collection of the muscle biopsies the samples will be stored under liquid nitrogen. The parameter evaluated in the muscles biopsies will be glycogen.

CONTACTS AND LOCATIONS:
Overall Officials: Per B Jeppesen, Prof., PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Dept of Clinical medicine, Aarhus C, Denmark